CLINICAL TRIAL: NCT00325442
Title: A 16-Week, International, Multicenter, Double-Blind, Randomized, Placebo-Controlled Comparison of the Efficacy and Safety of Oral UT-15C Sustained Release Tablets in Combination With an Endothelin Receptor Antagonist and/or a Phosphodiesterase-5 Inhibitor in Subjects With Pulmonary Arterial Hypertension
Brief Title: FREEDOM-C: Oral Treprostinil in Combination With an Endothelin Receptor Antagonist (ERA) and/or a Phosphodiesterase-5 (PDE-5) Inhibitor for the Treatment of Pulmonary Arterial Hypertension (PAH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDE-PH-301
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Active (Active Comparator): Subjects assigned to active therapy with UT-15C 0.25, 0.5, 1, or 5 mg oral tablets.
  Interventions: Drug: Oral treprostinil (UT-15C) sustained release tablets
- Placebo Arm (Placebo Comparator): Subjects assigned to placebo 0.25, 0.5, 1, or 5 mg oral tablets.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral treprostinil (UT-15C) sustained release tablets — UT-15C 0.25, 0.5, 1, or 5 mg oral tablets by mouth every 12 hours
  Arms: Active
Drug: Placebo — Placebo 0.25, 0.5, 1, or 5 mg oral tablets by mouth every 12 hours
  Arms: Placebo Arm

SUMMARY:
This study was an international, multi-center, randomized, double-blind, placebo-controlled study in subjects with PAH who were currently receiving approved therapy for their PAH (i.e., endothelin receptor antagonist and/or phosphodiesterase-5 inhibitor). Study visits occurred at 4 week intervals for 16 weeks; the key measure of efficacy was the 6-minute walk test. Study procedures included routine blood tests, medical history, physical exams, disease evaluation, and exercise tests. One optional substudy was also a part of FREEDOM-C at select centers - a hemodynamic substudy with a right heart catheterization at Baseline and Week 16.

Patients who completed all assessments for 16-weeks were also eligible to enter an open-label, extension phase study (FREEDOM - EXT).

ELIGIBILITY:
Inclusion Criteria:

* Between 12 and 70 years of age, inclusive.
* Body weight at least 45 kg (approximately 100 pounds).
* PAH that is either idiopathic/heritable (including PAH associated with appetite suppressant/toxin use); PAH associated with repaired congenital systemic-to-pulmonary shunts (repaired ≥ 5 years); PAH associated with collagen vascular disease; or PAH associated with HIV.
* Baseline 6-minute walk distance between 150 and 450 meters, inclusive.
* Currently receiving an approved endothelin receptor antagonist and/or an approved phosphodiesterase-5 inhibitor for at least 90 days and on a stable dose for at least the last 30 days.
* Previous testing (e.g., right heart catheterization, echocardiography) consistent with the diagnosis of PAH.
* Reliable and cooperative with protocol requirements.

Exclusion Criteria:

* Nursing or pregnant.
* Received a prostacyclin within the past 30 days.
* PAH due to conditions other than noted in the above inclusion criteria.
* History of uncontrolled sleep apnea, renal insufficiency, anemia, left sided heart disease, uncontrolled systemic hypertension, or parenchymal lung disease.
* Use of an investigational drug within 30 days of Baseline.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2006-10; Primary Completion 2008-09 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (72):
- United States (39):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Arizona Pulmonary Specialist, Phoenix, Arizona
  - University of Arizona Health Science Center, Tucson, Arizona
  - West Los Angeles VA Healthcare Center, Los Angeles, California
  - Stanford University, Pulmonary and Critical Care, Palo Alto, California
  - UC Davis Medical Center, Sacramento, California
  - University of California-San Francisco, San Francisco, California
  - Harbour-UCLA Medical Center, Torrance, California
  - The Children's Hospital, Aurora, Colorado
  - Pulmonary Hypertension Clinic, Aurora, Colorado
  - University of Chicago, Chicago, Illinois
  - University of Iowa Health Care, Iowa City, Iowa
  - Maine Medical Center, Portland, Maine
  - University of Maryland School of Medicine, Baltimore, Maryland
  - John's Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Hospital, St Louis, Missouri
  - Columbia Presbyterian Medical Center, New York, New York
  - Mary M Parkes Center for Asthma, Allergy and Pulmonary Care, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Legacy Clinic Northwest, Portland, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - Baylor College of Medicine, Pulmonary & Critical Care, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - Inova Transplant Center, Fairfax, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Heart Care Associates, Milwaukee, Wisconsin
- Australia (4):
  - St. Vincent's Hospital, Sydney, New South Wales
  - The Prince Charles Hospital, Brisbane
  - The Alfred Hospital, Melbourne
  - Royal Perth Hospital, Perth
- Austria (2):
  - Medizinische Universität Innsbruck, Innsbruck
  - Universitaet Wien, Vienna
- Belgium (2):
  - Hospital Erasme, Brussels
  - University Hospital Gasthuisberg, Leuven
- Canada (5):
  - Respiratory Research, Calgary, Alberta
  - Vancouver Coastal Health Respiratory Clinic, Vancouver, British Columbia
  - Lab London Health Sciences Center, London, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - SMBD Jewish General Hospital, Montreal, Quebec
- France (4):
  - Hospital Cavale Blanche, Brest
  - Hospital Antoine Beclere, Clamart
  - Hospital Claude Huriez, Lille
  - Hôpital Louis Pradel, Lyon
- Medizinische Hochschule Hannover, Hanover, Germany
- Mater Misericordiae University Hospital Ltd, Dublin, Ireland
- Israel (3):
  - Hadassah Ein-Kerem Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Tel Hashomer Medical Center, Ramat Gan
- Italy (2):
  - Universita degli Studi Bologna, Bologna
  - Universita "La Sapienza" Roma, Rome
- Hospital Vrije Universiteit, Amsterdam, Netherlands
- National Tuberculosis and Lung Disease Research Institute, Warsaw, Poland
- Spain (3):
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital Valle Hebron, Barcelona
  - Hospital 12 de Octubre, Madrid
- United Kingdom (4):
  - Papworth Hospital, Cambridge
  - Western Infirmary, Glasgow
  - Royal Free Hospital, London
  - Freeman Hospital, Newcastle

REFERENCES:
- [Derived] Lachant D, Raina A, Krishnan M, Sood N, Balasubramanian V, Barbera JA, Kiely DG, Lee D, Wu B, Hwang S, Seaman S, Broderick M, Elwing J. Efficacy and Safety of Oral Treprostinil in Patients with Pulmonary Arterial Hypertension on Background Monotherapy or Dual Therapy. Adv Ther. 2026 Feb 2. doi: 10.1007/s12325-026-03497-4. Online ahead of print. PMID 41627369
- [Derived] Tapson VF, Torres F, Kermeen F, Keogh AM, Allen RP, Frantz RP, Badesch DB, Frost AE, Shapiro SM, Laliberte K, Sigman J, Arneson C, Galie N. Oral treprostinil for the treatment of pulmonary arterial hypertension in patients on background endothelin receptor antagonist and/or phosphodiesterase type 5 inhibitor therapy (the FREEDOM-C study): a randomized controlled trial. Chest. 2012 Dec;142(6):1383-1390. doi: 10.1378/chest.11-2212. PMID 22628490

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 354 subjects were randomized with 350 subjects receiving a dose of study drug and subsequently analyzed from 20 October 2006 to 17 September 2008 at 70 sites across the United States, Canada, Europe, Israel, and Australia.
Groups:
- Placebo Arm: Subjects were randomly allocated to receive oral placebo twice daily.
- Active: Subjects in this arm were randomly allocated to receive oral treprostinil twice daily.
Period: Overall Study
Arm/Group | Placebo Arm | Active
Started | 176 | 174
Completed | 167 | 153
Not Completed | 9 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Arm | Active | Total
Number analyzed (Participants) | 176 | 174 | 350
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 3 | 8
  Between 18 and 65 years | 149 | 151 | 300
  >=65 years | 22 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (13.3) | 51.1 (12.3) | 50.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 148 | 288
  Male | 36 | 26 | 62
Distance Traversed (meters) During Six Minute Walk Test at Baseline [Mean (Standard Deviation); unit: meters] | 345.4 (75.5) | 346.1 (71.4) | 345.7 (73.4)
Baseline WHO Functional Classification [Number; unit: participants] — Class I: PH without limitation of physical activity (PA); no undue dyspnea or fatigue, chest pain, or near syncope.
  Class II: PH resulting in slight limitation of PA; comfortable at rest; ordinary PA causes undue dyspnea or fatigue, chest pain or near syncope.
  Class III: PH resulting in marked limitation of PA; comfortable at rest; ordinary PA causes undue dyspnea or fatigue, chest pain, or near syncope.
  Class IV: PH with inability to carry out any PA without symptoms and signs of right heart failure. Dyspnea and/or fatigue may be present at rest. Discomfort is increased by any PA.
  participants
    WHO Functional Class I | 1 | 2 | 3
    WHO Functional Class II | 31 | 41 | 72
    WHO Functional Class III | 139 | 127 | 266
    WHO Functional Class IV | 5 | 4 | 9
PAH Etiology [Number; unit: participants]
  Idiopathic / familial PAH | 119 | 113 | 232
  PAH associated with collagen vasular disease | 43 | 49 | 92
  PAH associated wtih congenital heart defect | 11 | 11 | 22
  PAH associated with HIV infection | 3 | 1 | 4
Background PAH Therapy [Number; unit: participants]
  ERA | 51 | 55 | 106
  PDE5-I | 43 | 45 | 88
  ERA and PDE5-I | 82 | 74 | 156

OUTCOME MEASURES:

1. Primary Outcome: Six Minute Walk Distance (6MWD)
Description: Placebo corrected change in six minute walk distance (6MWD) from Baseline to Week 16, correlates with the historical clinical standard for assessing patient functional status in the treatment of PAH and is considered an objective measure of patient functional status by the American Thoracic Society (ATS).
  The six minute walk test was to be conducted 3 to 6 hours after the previous dose of study drug.
Time Frame: Baseline and 16 Weeks
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 176 | 174
meters
  6MWD at Baseline | 362.5 [302.0 to 400.0] | 362.5 [304.0 to 397.0]
  6MWD at Week 16 | 367.0 [283.0 to 420.5] | 381.0 [323.0 to 420.0]
  Change in 6MWD from Baseline to Week 16 | 4.8 [-22.0 to 35.5] | 14.5 [-10.0 to 47.0]
Statistical Analysis 1: Comparison: Placebo Arm vs Active; Change in 6MWD from Baseline to Week 16; Test type: Superiority or Other; p = 0.072, ANCOVA; Hodges-Lehmann = 11.0, 95% CI 2-sided [0 to 22]

2. Secondary Outcome: Borg Dyspnea Score
Description: The Borg dyspnea score is a 10-point scale rating the maximum level of dyspnea experienced during the 6-minute walk test. The Borg dyspnea score was assessed immediately following the 6-minute walk test. Scores ranged from 0 (for no shortness of breath) to 10 (for greatest shortness of breath ever experienced).
Time Frame: Baseline and 16 Weeks
Population: One subject in the placebo arm did not have a Baseline Borg score value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 175 | 174
units on a scale
  Borg dyspnea score at Baseline | 4.26 (2.25) | 4.22 (2.24)
  Borg dyspnea score at Week 16 | 4.64 (2.62) | 4.18 (2.59)
  Change in Borg dyspnea score from BL to Wk 16 | 0.38 (2.06) | -0.03 (2.13)
Statistical Analysis 1: Comparison: Placebo Arm vs Active; Change in Borg dyspnea score from Baseline to Week 16; Test type: Superiority or Other; p = 0.062, Wilcoxon rank-sum test; Hodges-Lehmann (H-L) = 0.0, 95% CI 2-sided [-1.0 to 0.0]

3. Secondary Outcome: Clinical Worsening Assessment
Description: Definition of clinical worsening required one of the following:
  1. Death (all causes excluding accident)
  2. Transplantation or atrial septostomy
  3. Clinical deterioration as defined by:
     1. Hospitalization as a result of PAH, or
     2. ≥ 20% decrease in 6-minute walk distance from Baseline (or too ill to walk) and a decrease in WHO functional class And
     3. Initiation of new PAH specific therapy (i.e., ERA, PDE5I, prostacyclin).
Time Frame: Baseline and 16 Weeks
Measure: Number; unit: participants
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 176 | 174
participants | 12 | 8
Statistical Analysis 1: Comparison: Placebo Arm vs Active; Test type: Superiority or Other; p = 0.491, Fisher Exact

4. Secondary Outcome: Dyspnea-Fatigue Index
Description: The dyspnea-fatigue index has three components, each rated on a scale of 0 to 4, for the magnitude of the task that evokes dyspnea or fatigue, the magnitude of the pace (or effort) with which the task is performed and the associated functional impairment in general activities. The ratings for each component were added to form an aggregate score, which could range from 0, for the worst condition, to 12, for the best.
Time Frame: Baseline and 16 Weeks
Population: Five subjects in the placebo arm and three subjects in the active arm did not have a Baseline dypsnea-fatigue index score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 171 | 171
units on a scale
  Dyspnea-fatigue index at Baseline | 5.5 (2.2) | 5.7 (2.1)
  Dyspnea-fatigue index at Week 16 | 5.1 (2.5) | 5.7 (2.5)
  Change in dyspnea-fatigue index from BL to Wk 16 | -0.4 (1.9) | 0.0 (1.9)
Statistical Analysis 1: Comparison: Placebo Arm vs Active; Change in dyspnea-fatigue index from Baseline to Week 16; Test type: Superiority or Other; p = 0.011, Wilcoxon sum-rank test; Hodges-Lehmann (H-L) = 0.0, 95% CI 2-sided [0.0 to 1.0]

5. Secondary Outcome: World Health Organization Functional Classification for PAH
Description: Class I: Patients with pulmonary hypertension but without resulting limitation of physical activity. Ordinary physical activity does not cause undue dyspnea or fatigue, chest pain, or near syncope.
  Class II: Patients with pulmonary hypertension resulting in slight limitation of physical activity. These patients are comfortable at rest, but ordinary physical activity causes undue dyspnea or fatigue, chest pain or near syncope.
  Class III: Patients with pulmonary hypertension resulting in marked limitation of physical activity. They are comfortable at rest. Ordinary activity causes undue dyspnea or fatigue, chest pain, or near syncope.
  Class IV: Patients with pulmonary hypertension with inability to carry out any physical activity without symptoms. These patients manifest signs of right heart failure. Dyspnea and/or fatigue may be present even at rest. Discomfort is increased by any physical activity.
Time Frame: Week 16
Measure: Number; unit: participants
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 176 | 174
participants
  WHO Class I | 1 | 2
  WHO Class II | 48 | 58
  WHO Class III | 114 | 103
  WHO Class IV | 13 | 11

6. Secondary Outcome: Six Minute Walk Distance (6MWD)
Description: Placebo corrected change in six minute walk distance (6MWD) from Baseline to Week 12, correlates with the historical clinical standard for assessing patient functional status in the treatment of PAH and is considered an objective measure of patient functional status by the American Thoracic Society (ATS).
  The six minute walk test was to be conducted 3 to 6 hours after the previous dose of study drug.
Time Frame: Baseline and 12 weeks
Measure: Median (Full Range); unit: meters
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 176 | 174
meters
  6MWD at Baseline | 362.5 [302.0 to 400.0] | 362.5 [304.0 to 397.0]
  6MWD at Week 12 | 366.4 [280.5 to 424.0] | 378.0 [320.0 to 425.0]
  Change in 6MWD from Baseline to Week 12 | 5.8 [-23.5 to 29.5] | 16.5 [-15.0 to 51.0]
Statistical Analysis 1: Comparison: Placebo Arm vs Active; Change in 6MWD from Baseline to Week 12; Test type: Superiority or Other; p = 0.015, ANCOVA; Hodges-Lehmann (H-L) = 13.0, 95% CI 2-sided [3.0 to 23.0]

7. Secondary Outcome: Six Minute Walk Distance (6MWD)
Description: Placebo corrected change in six minute walk distance (6MWD) from Baseline to Week 8, correlates with the historical clinical standard for assessing patient functional status in the treatment of PAH and is considered an objective measure of patient functional status by the American Thoracic Society (ATS).
  The six minute walk test was to be conducted 3 to 6 hours after the previous dose of study drug.
Time Frame: Baseline and 8 weeks
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 176 | 174
meters
  6MWD at Baseline | 362.5 [302.0 to 400.0] | 362.5 [304.0 to 397.0]
  6MWD at Week 8 | 368.5 [294.5 to 416.0] | 379.0 [310.0 to 415.0]
  Change in 6MWD from Baseline to Week 8 | 7.0 [-22.0 to 30.5] | 15.0 [-9.0 to 42.0]
Statistical Analysis 1: Comparison: Placebo Arm vs Active; Change in 6MWD from Baseline to Week 8; Test type: Superiority or Other; p = 0.051, ANCOVA; Hodges-Lehmann = 9.0, 95% CI 2-sided [0.0 to 18.0]

8. Secondary Outcome: Six Minute Walk Distance (6MWD)
Description: Placebo corrected change in six minute walk distance (6MWD) from Baseline to Week 4, correlates with the historical clinical standard for assessing patient functional status in the treatment of PAH and is considered an objective measure of patient functional status by the American Thoracic Society (ATS).
  The six minute walk test was to be conducted 3 to 6 hours after the previous dose of study drug.
Time Frame: Baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 176 | 174
meters
  6MWD at Baseline | 362.5 [302.0 to 400.0] | 362.5 [304.0 to 397.0]
  6MWD at Week 4 | 363.0 [299.0 to 410.5] | 370.5 [312.0 to 410]
  Change in 6MWD from Baseline to Week 4 | 2.1 [-17.5 to 24.5] | 5.5 [-8.0 to 31.0]
Statistical Analysis 1: Comparison: Placebo Arm vs Active; Change in 6MWD from Baseline to Week 4; Test type: Superiority or Other; p = 0.238, ANCOVA; Hodges-Lehmann ( H-L) = 4, 95% CI 2-sided [-2.4 to 12.0]

9. Post Hoc Outcome: Six Minute Walk Distance (6MWD) by Baseline 6MWD Quartiles: Quartile 1 (126-302 Meters)
Time Frame: Baseline and 16 weeks
Population: The study population was divided into quartiles by Baseline 6MWD. The subjects in this subgroup were in quartile 1 (126 - 302 meters).
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 45 | 43
meters
  6MWD at Baseline | 247.0 [191.0 to 288.0] | 255.0 [204.0 to 289.0]
  6MWD at Week 16 | 241.0 [141.0 to 286.0] | 265.0 [189.0 to 325.0]
  Change in 6MWD from Baseline to Week 16 | -5.6 [-39.0 to 16.0] | 17.0 [-13.0 to 43.0]
Statistical Analysis 1: Comparison: Placebo Arm vs Active; Change in 6MWD from Baseline to Week 16; Test type: Superiority or Other; p = 0.121, ANCOVA; Hodges-Lehmann (H-L) = 24, 95% CI 2-sided [0 to 45]

10. Post Hoc Outcome: Six Minute Walk Distance (6MWD) by Baseline 6MWD Quartile: Quartile 2 (303 - 362 Meters)
Time Frame: Baseline and 16 weeks
Population: The study population was divided into quartiles by Baseline 6MWD. The subjects in this subgroup were in quartile 2 (303 - 362 meters).
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 43 | 44
meters
  6MWD at Baseline | 332.0 [323.0 to 354.0] | 339.0 [323.5 to 350.5]
  6MWD at Week 16 | 348.0 [300.0 to 376.0] | 359.0 [329.5 to 400.5]
  Change in 6MWD from Baseline to Week 16 | 12.0 [-22.0 to 37.0] | 17.0 [-0.4 to 53.0]
Statistical Analysis 1: Comparison: Placebo Arm vs Active; Change in 6MWD from Baseline to Week 16; Test type: Superiority or Other; p = 0.069, ANCOVA; Hodges-Lehmann (H-L) = 15, 95% CI 2-sided [-7 to 41]

11. Post Hoc Outcome: Six Minute Walk Distance (6MWD) by Baseline 6MWD Quartile: Quartile 3 (363 - 397 Meters)
Time Frame: Baseline and 16 weeks
Population: The study population was divided into quartiles by Baseline 6MWD. The subjects in this subgroup were in quartile 3 (363 - 397 meters).
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 42 | 45
meters
  6MWD at Baseline | 385.0 [378.0 to 390.0] | 383.0 [376.0 to 390.0]
  6MWD at Week 16 | 388.0 [358.0 to 429.0] | 396.0 [370.0 to 417.0]
  Change in 6MWD from Baseline to Week 16 | 6.5 [-22.0 to 43.0] | 13.0 [-8.0 to 44.0]
Statistical Analysis 1: Comparison: Placebo Arm vs Active; Change in 6MWD from Baseline to Week 16; Test type: Superiority or Other; p = 0.889, ANCOVA; Hodges-Lehmann (H-L) = 4, 95% CI 2-sided [-15 to 24]

12. Post Hoc Outcome: Six Minute Walk Distance (6MWD) by Baseline 6MWD Quartile: Quartile 4 (398 - 450 Meters)
Time Frame: Baseline and 16 weeks
Population: The study population was divided into quartiles by Baseline 6MWD. The subjects in this subgroup were in quartile 4 (398 - 450 meters).
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 46 | 42
meters
  6MWD at Baseline | 425.5 [410.0 to 440.0] | 425.0 [412.0 to 430.0]
  6MWD at Week 16 | 442.0 [411.0 to 468.0] | 438.5 [395.0 to 483.0]
  Change in 6MWD from Baseline to Week 16 | 15.0 [-6.0 to 49.0] | 15.0 [-20.0 to 59.0]
Statistical Analysis 1: Comparison: Placebo Arm vs Active; Change in 6MWD from Baseline to Week 16; Test type: Superiority or Other; p = 0.966, ANCOVA; Hodges-Lehmann (H-L) = 0, 95% CI 2-sided [-23 to 24]

13. Post Hoc Outcome: Change in Six Minute Walk Distance (6MWD) From Baseline in Subjects Who Received Oral Treprostinil by Last Study Drug Dose and Reason for Discontinuation
Description: In general, the dose of study drug was increased in 0.5 mg increments every 3 days, in the absence of dose-limiting drug-related AEs, to ensure the subject received the optimal clinical dose throughout the study.
Time Frame: Baseline and 16 weeks
Population: Of 174 subjects randomized to receive oral treprostinil, 153 subjects who completed the study and 6 additional subjects who did not complete the study but discontinued the study due to adverse events were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: meters
Groups:
- Less Than 1 mg or Discontinuation Due to Adverse Events: Subjects in this group received less than or equal to 1 mg oral treprostinil twice daily or discontinued treatment due to adverse events.
- 1.25 - 3.25 mg: Subjects in this group recieved 1.25 to 3.25 mg oral treprostinil twice daily.
- 3.5 - 16 mg: Subjects in this group received 3.5 to 16 mg oral treprostinil twice daily.
Arm/Group | Less Than 1 mg or Discontinuation Due to Adverse Events | 1.25 - 3.25 mg | 3.5 - 16 mg
Number analyzed (Participants) | 58 | 49 | 52
meters | 3.8 [-8.0 to 26.0] | 18.0 [-3.0 to 56.0] | 34.0 [3.0 to 52.0]

14. Post Hoc Outcome: Six Minute Walk Distance (6MWD) by Lowest Dose Strength Available at Randomization: Smallest Dose Available 1 mg
Time Frame: Baseline and 16 weeks
Population: The subjects in this subgroup had a minimum tablet strength of 1 mg for initiation of study drug dosing and dose titration.
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 51 | 51
meters
  6MWD at Baseline | 348.0 [282.0 to 385.0] | 349.0 [311.0 to 380.0]
  6MWD at Week 16 | 350.0 [243.0 to 431.0] | 379.0 [324.7 to 405.0]
  Change in 6MWD from Baseline to Week 16 | 15.0 [-26.0 to 55.0] | 22.0 [5.0 to 45.0]
Statistical Analysis 1: Comparison: Placebo Arm vs Active; Change in 6MWD from Baseline to Week 16; Test type: Superiority or Other; p = 0.853, ANCOVA; Hodges-Lehmann (H-L) = 5, 95% CI 2-sided [-16 to 28]

15. Post Hoc Outcome: Six Minute Walk Distance (6MWD) by Lowest Study Drug Dose Strength Available at Randomizaiton: Dose Strength 0.5 mg
Time Frame: Baseline and 16 weeks
Population: The subjects in this subgroup had a minimum tablet strength of 0.5 mg for initiation of study drug dosing and dose titration.
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 99 | 100
meters
  6MWD at Baseline | 366.0 [302.0 to 410.0] | 370.0 [297.0 to 411.0]
  6MWD at Week 16 | 370.0 [283.0 to 430.0] | 375.5 [301.0 to 439.5]
  Change in 6MWD from Baseline to Week 16 | 7.0 [-19.0 to 30.0] | 7.0 [-19.0 to 46.5]
Statistical Analysis 1: Comparison: Placebo Arm vs Active; Change in 6MWD from Baseline to Week 16; Test type: Superiority or Other; p = 0.327, ANCOVA; Hodges-Lehmann (H-L) = 7, 95% CI 2-sided [-7 to 21]

16. Post Hoc Outcome: Six Minute Walk Distance (6MWD) by Lowest Study Drug Dose Strength Available at Randomization: Study Drug Dose 0.25 mg
Time Frame: Baseline and 16 weeks
Population: The subjects in this subgroup had a minimum tablet strength of 0.25 mg for initiation of study drug dosing and dose titration.
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 26 | 23
meters
  6MWD at Baseline | 374.0 [319.0 to 408.0] | 384.0 [306.0 to 405.0]
  6MWD at Week 16 | 374.0 [320.0 to 399.0] | 398.0 [340.0 to 438.0]
  Change in 6MWD from Baseline to Week 16 | -1.0 [-30.0 to 12.0] | 21.0 [-7.0 to 78.0]
Statistical Analysis 1: Comparison: Placebo Arm vs Active; Change in 6MWD from Baseline to Week 16; Test type: Superiority or Other; p = 0.085, ANCOVA; Hodges-Lehmann (H-L) = 29.5, 95% CI 2-sided [1 to 73]

17. Post Hoc Outcome: Six Minute Walk Distance (6MWD) by Background PAH Therapy: ERA
Time Frame: Baseline and 16 weeks
Population: The subjects in this subgroup were receiving treatment with an ERA for 90 days or greater at the time of randomization.
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 51 | 55
meters
  6MWD at Baseline | 382.0 [325.0 to 403.0] | 372.0 [325.0 to 398.0]
  6MWD at Week 16 | 377.0 [303.0 to 423.0] | 385.0 [306.4 to 422.0]
  Change in 6MWD from Baseline to Week 16 | -3.0 [-22.0 to 30.0] | 4.0 [-16.0 to 40.0]
Statistical Analysis 1: Comparison: Placebo Arm vs Active; Change in 6MWD from Baseline to Week 16; Test type: Superiority or Other; p = 0.615, ANCOVA; Hodges-Lehmann (H-L) = 5, 95% CI 2-sided [-12 to 24]

18. Post Hoc Outcome: Six Minute Walk Distance (6MWD) by Background PAH Therapy: PDE5-I
Time Frame: Baseline and 16 weeks
Population: The subjects in this subgroup were receiving treatment with a PDE5-I for 90 days or greater at the time of randomization.
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 43 | 45
meters
  6MWD at Baseline | 360.0 [302.0 to 397.0] | 348.0 [296.0 to 390.0]
  6MWD at Week 16 | 357.0 [318.0 to 424.0] | 373.0 [307.0 to 411.0]
  Change in 6MWD from Baseline to Week 16 | 8.0 [-31.0 to 47.0] | 23.0 [-3.0 to 47.0]
Statistical Analysis 1: Comparison: Placebo Arm vs Active; Change in 6MWD from Baseline to Week 16; Test type: Superiority or Other; p = 0.230, ANCOVA; Hodges-Lehmann (H-L) = 17, 95% CI 2-sided [-6 to 40]

19. Post Hoc Outcome: Six Minute Walk Distance (6MWD) by Background PAH Therapy: ERA and PDE5-I
Time Frame: Baseline and 16 weeks
Population: The subjects in this subgroup were receiving treatment with an ERA and PDE5-I for 90 days or greater at the time of randomization.
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 82 | 74
meters
  6MWD at Baseline | 351.5 [290.0 to 400.0] | 358.5 [300.0 to 412.0]
  6MWD at Week 16 | 359.2 [243.0 to 418.0] | 381.0 [325.0 to 425.0]
  Change in 6MWD from Baseline to Week 16 | 8.0 [-20.0 to 35.0] | 14.5 [-13.0 to 47.0]
Statistical Analysis 1: Comparison: Placebo Arm vs Active; Change in 6MWD from Baseline to Week 16; Test type: Superiority or Other; p = 0.209, ANCOVA; Hodges-Lehmann (H-L) = 10, 95% CI 2-sided [-6 to 28]

20. Secondary Outcome: Change in Symptoms of PAH From Baseline to Week 16
Description: Defined symptoms of PAH including fatigue, dyspnea, edema, dizziness, syncope, chest pain, and orthopnea were assessed at Baseline prior to starting study drug and during the Treatment Phase at Week 16. Severity grade values (i.e., 0, 1, 2, or 3 in increasing severity) were assigned for each symptom. The outcome data describes the change in severity values from Baseline to Week 16 for each defined symptom of PAH.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Arm | Active
Number analyzed (Participants) | 176 | 174
units on a scale
  Change in fatigue symptoms | 0.0 (0.0) | 0.01 (0.10)
  Change in dypsnea symptoms | 0.00 (0.00) | -0.01 (0.09)
  Change in edema symptoms | 0.00 (0.00) | -0.06 (0.10)
  Change in dizziness symptoms | 0.00 (0.00) | -0.16 (0.11)
  Change in syncope symptoms | 0.00 (0.00) | -0.10 (0.09)
  Change in chest pain symptoms | 0.00 (0.00) | -0.09 (0.11)
  Change in orthopnea symptoms | 0.00 (0.00) | -0.20 (0.10)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout the 16 week study which was conducted between October 2006 and September 2008.
Arm/Group | Placebo Arm | Active
Serious Adverse Events (participants affected / at risk) | 33/176 | 32/174
Other Adverse Events (participants affected / at risk) | 157/176 | 173/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (N=176) | Active (N=174)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 9 (9)
right ventricular failure (Cardiac disorders) | 2 (2) | 6 (7)
syncope (General disorders) | 3 (3) | 2 (4)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
atrial flutter (Cardiac disorders) | 1 (1) | 2 (2)
renal failure acute (Renal and urinary disorders) | 0 (0) | 3 (4)
chest pain (Cardiac disorders) | 2 (2) | 0 (0)
hypotension (Vascular disorders) | 2 (2) | 0 (0)
lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
aortic stenosis (Cardiac disorders) | 0 (0) | 1 (1)
bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
diarrhea hemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
epistaxis (Vascular disorders) | 1 (1) | 0 (0)
fluid overload (Vascular disorders) | 1 (1) | 0 (0)
fluid retention (Vascular disorders) | 1 (1) | 0 (0)
gastroenteritis viral (Gastrointestinal disorders) | 1 (1) | 0 (0)
hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0)
hyperparathyroidism secondary (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hypersensitivity (General disorders) | 1 (1) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
infection (Infections and infestations) | 1 (1) | 0 (0)
international normalized ratio increased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
iron deficiency anemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
liver function test abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
low cardiac output syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pericarditis constrictive (Cardiac disorders) | 1 (1) | 0 (0)
pulmonary hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
pyrexia (Infections and infestations) | 1 (1) | 0 (0)
spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
subarachnoid hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
subdural hematoma (Nervous system disorders) | 1 (1) | 0 (0)
suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
tibia fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
large intestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
central line infection (Infections and infestations) | 0 (0) | 1 (1)
hepatic enzyme increased (Hepatobiliary disorders) | 0 (0) | 1 (1)
streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (N=176) | Active (N=174)
headache (Nervous system disorders) | 65 (69) | 150 (164)
nausea (Gastrointestinal disorders) | 60 (65) | 112 (126)
diarrhea (Gastrointestinal disorders) | 48 (49) | 106 (115)
flushing (Vascular disorders) | 27 (28) | 85 (87)
pain in jaw (Musculoskeletal and connective tissue disorders) | 21 (22) | 75 (77)
vomiting (Gastrointestinal disorders) | 14 (18) | 76 (82)
pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (17) | 54 (62)
dizziness (Ear and labyrinth disorders) | 28 (33) | 30 (33)
fatigue (General disorders) | 17 (18) | 25 (25)
edema peripheral (Vascular disorders) | 17 (19) | 15 (15)
myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 24 (26)
nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 13 (14)
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 11 (11)
chest pain (Cardiac disorders) | 14 (15) | 12 (12)
palpitations (Cardiac disorders) | 9 (9) | 17 (18)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 13 (14)
back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 13 (13)
pain (General disorders) | 6 (7) | 17 (17)
arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 18 (19)
cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 11 (11)
insomnia (Nervous system disorders) | 7 (7) | 15 (15)
abdominal distention (Vascular disorders) | 10 (10) | 11 (11)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 11 (11)
pulmonary arterial hypertension (Vascular disorders) | 11 (12) | 10 (10)
rash (Skin and subcutaneous tissue disorders) | 8 (8) | 10 (11)
syncope (General disorders) | 11 (14) | 7 (9)
constipation (Gastrointestinal disorders) | 8 (8) | 9 (9)
dyspepsia (Gastrointestinal disorders) | 8 (10) | 9 (9)
abdominal pain upper (Musculoskeletal and connective tissue disorders) | 8 (8) | 8 (8)
epistaxis (Vascular disorders) | 9 (10) | 7 (7)
decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 13 (13)
abdominal pain (General disorders) | 5 (5) | 8 (8)
anxiety (Psychiatric disorders) | 4 (4) | 8 (10)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 9 (9)
oropharyngeal pain (General disorders) | 8 (8) | 3 (3)
migraine (Nervous system disorders) | 0 (0) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the results of this trial must be consistent with the United Therapeutics publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.